CLINICAL TRIAL: NCT05554926
Title: A Phase 1, Open-label Study of the Absorption, Metabolism, and Excretion of [4-14C] AEF0117 Following a Single Oral Dose in Healthy Male Subjects
Brief Title: Study of [4-14C] AEF0117 Following a Single Oral Dose in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aelis Farma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AEF0117-106
Record Dates: First submitted 2022-09-22; First posted 2022-09-26 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Marijuana Abuse
Keywords: AEF0117
MeSH Terms: conditions — Marijuana Abuse

STUDY DESIGN:
Intervention Model Description: Up to 8 subjects will be enrolled to ensure that 6 subjects complete the study. Subjects will be admitted into the study site on Day -1.
  On the morning of Day 1, all subjects will receive a single oral dose of 2 mg containing approximately 100 μCi of [4-14C]AEF0117 approximately 1 hour after completion of a low-fat breakfast.
  Subjects will reside at the study site from Day -1 through Day 28 and will be discharged on Day 28
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- [4-14C] AEF0117 (Experimental): Potential subjects will be screened to assess their eligibility to enter the study within 28 days prior to the dose administration. Up to 8 subjects will be enrolled to ensure that 6 subjects complete the study. Subjects will be admitted into the study site on Day -1. On the morning of Day 1, all subjects will receive a single oral dose of 2 mg containing approximately 100 μCi of [4-14C]AEF0117 approximately 1 hour after completion of a low-fat breakfast
  Interventions: Drug: AEF0117

INTERVENTIONS:
Drug: AEF0117 — 2 mg AEF0117 containing approximately 100 μCi of [4-14C]AEF0117
  Other Names: 3ß-(4-methoxybenzykoxy)pregn-5-en-20-one t)

SUMMARY:
Cannabis use is increasing and will only further escalate with legalization of recreational and medical cannabis use in western countries , with a prevalence greater than 30 % in the US and most European countries for individuals between 16 and 24 years of age. Approximately 9 % of those who use cannabis will become addicted. The number goes up to about 1 in 6 among those who start using cannabis as teenagers and to 25 to 50 % among those who smoke cannabis daily. The consequences of cannabis abuse in the most prone population (14-25 years of age) are extremely serious, and may include addiction, altered brain development, poorer educational outcomes, cognitive impairment, lower income, greater welfare dependence, unemployment and lower relationship and life satisfaction. There are no available pharmacological treatments of cannabis use disorder (CUD). Thus, the development of safe and effective medications for the treatment of CUD is an urgent public health priority.

The preclinical efficacy and available ADMET (Administration, Distribution, Metabolism, Elimination and Toxicology) in animal and human data suggest that AEF0117, an investigational new study drug, could constitute a very efficacious and safe treatment for cannabis abuse disorders. The purpose of this research is to study how AEF0117 influences the subjective effects of cannabis in subjects with CUD. AEF0117 acts in the same parts of the brain as THC (tetrahydrocannabinol), the active ingredient of marijuana, and may temporarily alter some of cannabis's effects.

This will be a Phase 1, open-label, nonrandomized, single-dose study in healthy male subjects. Potential subjects will be screened to assess their eligibility to enter the study within 28 days prior to the dose administration. Subjects will be admitted into the study site on Day 1. On the morning of Day 1, all subjects will receive a single oral dose of 2 mg containing approximately 100 μCi of [4-14C]AEF0117 approximately 1 hour after completion of a low fat breakfast.

DETAILED DESCRIPTION:
Cannabis use is increasing and will only further escalate with legalization of recreational and medical cannabis use in western countries , with a prevalence greater than 30 % in the US and most European countries for individuals between 16 and 24 years of age. Approximately 9 % of those who use cannabis will become addicted. The number goes up to about 1 in 6 among those who start using cannabis as teenagers and to 25 to 50 % among those who smoke cannabis daily. The consequences of cannabis abuse in the most prone population (14-25 years of age) are extremely serious, and may include addiction, altered brain development, poorer educational outcomes, cognitive impairment, lower income, greater welfare dependence, unemployment and lower relationship and life satisfaction. There are no available pharmacological treatments of cannabis use disorder (CUD). Thus, the development of safe and effective medications for the treatment of CUD is an urgent public health priority.

The preclinical efficacy and available ADMET (Administration, Distribution, Metabolism, Elimination and Toxicology) in animal and human data suggest that AEF0117, an investigational new study drug, could constitute a very efficacious and safe treatment for cannabis abuse disorders. The purpose of this research is to study how AEF0117 influences the subjective effects of cannabis in subjects with CUD. AEF0117 acts in the same parts of the brain as THC (tetrahydrocannabinol), the active ingredient of marijuana, and may temporarily alter some of cannabis's effects.

The safety and tolerability of AE0117 has been demonstrated in the clinical studies conducted to date.

The purpose of this study is to determine the absorption, metabolism, and excretion of [4 14C]AEF0117 and to characterize and determine the metabolites present in plasma, urine, and, where possible, feces in healthy male subjects following a single oral administration. Knowledge of the metabolism and excretion of parent drug and its metabolites is useful for evaluating the Metabolites in Safety Testing requirements elucidated in the Food and Drug Administration (FDA) Guidance and International Conference on Harmonisation (ICH) M3 and the likelihood of effects of renal or hepatic impairment on the disposition of AEF0117 and the likelihood for drug-drug interactions with AEF0117.

This will be a Phase 1, open-label, nonrandomized, single dose study in healthy male subjects.

Potential subjects will be screened to assess their eligibility to enter the study within 28 days prior to the dose administration. Up to 8 subjects will be enrolled to ensure that 6 subjects complete the study. Subjects will be admitted into the study site on Day 1. On the morning of Day 1, all subjects will receive a single oral dose of 2 mg containing approximately 100 μCi of [4-14C]AEF0117 approximately 1 hour after completion of a low fat breakfast.

Subjects will reside at the study site from Day -1 through Day 28 and will be discharged on Day 28. If the following criteria are not met by Day 28, subjects will continue study participation and will be asked to return for a residential visit on Day 35 to allow for continuation of the 24-hour collection (urine, blood, and feces) for total radioactivity:

* plasma radioactivity levels below the limit of quantitation for 2 consecutive collections,
* ≥90% mass balance recovery, and
* ≤1% of the total radioactive dose is recovered in combined excreta (urine and feces) in 2 consecutive 24-hour periods.

If the following criteria are not met at the Day 35 visit, then the subjects will be required to come back on Day 42 to allow for continuation of the 24-hour collection (urine, blood, and feces) for total radioactivity:

* plasma radioactivity levels below the limit of quantitation for 2 consecutivecollections, and
* ≤1% of the total radioactive dose is recovered in combined excreta (urine and feces) in 24-hour period.

Subjects will be discharged from the study at the latest discharge day of Day 43, unlessotherwise agreed upon by the sponsor and investigator.

Up to 8 subjects will be enrolled to ensure that 6 subjects complete the study.

ELIGIBILITY:
Inclusion Criteria:

1. Males, of any race, between 18 and 65 years of age, inclusive, at screening.
2. Body mass index between 18.0 and 30.0 kg/m2, inclusive.
3. In good health, determined by no clinically significant findings from medical history,12-lead electrocardiogram (ECG), vital signs measurements, and clinical laboratory evaluations (congenital nonhemolytic hyperbilirubinemia [eg, suspicion of Gilbert's syndrome based on total and direct bilirubin] is not acceptable) at screening and check-in and from the physical examination at check-in, as assessed by the investigator (or designee).
4. Males will agree to use contraception
5. Able to comprehend and willing to sign an ICF and to abide by the study restrictions.
6. History of a minimum of one bowel movement per day.

Exclusion Criteria:

Medical conditions

1. Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder, as determined by the investigator (or designee).
2. History of significant hypersensitivity, intolerance, or allergy to corn products/oil, or allergy to any drug compound, food, or other substance, unless approved by the investigator (or designee).
3. History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs (uncomplicated appendectomy and hernia repair will be allowed). Cholecystectomy is not allowed.
4. Confirmed vital signs measurements below:

   * systolic blood pressure >140 or <90 mmHg, systolic blood pressure >160 or <90 mmHg for male volunteers between 60 and 65 years old
   * diastolic blood pressure >90 or <50 mmHg, and
   * pulse rate >100 or <40 beats per minute. Minor deviations from the normal range may be allowed if deemed by the investigator to have no clinical significance, after discussion with medical monitor.
5. Positive hepatitis panel and/or reactive human immunodeficiency virus test
6. Positive coronavirus disease 2019 (COVID-19) test less than 30 days prior to screening and/or experiencing symptoms.

   Prior/concomitant therapy
7. Administration of a COVID-19 vaccine in the past 30 days prior to dosing.
8. Use or intend to use any medications/products known to alter drug absorption, metabolism, or elimination processes, including St. John's wort, and/or use or intend to use any drugs known to induce or inhibit CYP isozymes, within 30 days prior to check-in, unless deemed acceptable by the investigator (or designee) and accepted by sponsor's medical monitor.
9. Use or intend to use any prescription medications/products within 14 days prior to check-in, and any medication with an elimination half-life of >60 hours (time since last dose of at least 6 times the elimination half-life), unless deemed acceptable by the investigator (or designee) and with consultation with sponsor's medical monitor.
10. Use or intend to use slow-release medications/products considered to still be activewithin 14 days prior to check-in, unless deemed acceptable by the investigator (or designee) and accepted by sponsor's medical monitor.
11. Use or intend to use any nonprescription medications/products including vitamins,minerals, and phytotherapeutic/herbal/plant-derived preparations within 7 days priorto check-in, unless deemed acceptable by the investigator (or designee) and with consultation with sponsor's medical monitor.

    Prior/concurrent clinical study experience
12. Participation in a clinical study involving administration of an investigational drug (new chemical entity) in the past 30 days or 5 half-lives (if known) prior to dosing, and if the elimination half-life is >60 hours (time since last dose of at least 6 times the elimination half-life), following agreement between investigator (or designee) and sponsor's medical monitor.
13. Subjects who have participated in more than 3 radiolabeled drug studies in the last 12 months (previous study to be at least 4 months prior to check-in to the study site where exposures are known to the investigator or 6 months prior to check-in to the study site for a radiolabeled drug study where exposures are not known to the investigator). The total 12-month exposure from this study and a maximum of 2 other previous radiolabeled studies within 4 to 12 months prior to this study will be within the Code of Federal Regulations (CFR) recommended levels considered safe, per the US Title 21 CFR 361.1.
14. Have previously completed or withdrawn from this study or any other study investigating AEF0117 and have previously received AEF0117.

    Diet and lifestyle
15. Alcohol consumption of >21 units per week for males. One unit of alcohol equals 12 oz (360 mL) beer, 1½ oz (45 mL) liquor, or 5 oz (150 mL) wine.
16. Positive urine drug screen at screening or check-in or positive urine alcohol test result at check-in.
17. History of alcoholism or drug/chemical abuse (as defined by the current Diagnostic and Statistical Manual of Mental Disorders) within 2 years prior to check-in.
18. Use of tobacco- or nicotine-containing products within 3 months prior to check-in or positive cotinine at screening or check-in.

    Other exclusions
19. Receipt of blood products within 2 months prior to check-in.
20. Donation of blood from 3 months prior to screening, plasma from 2 weeks prior to screening, or platelets from 6 weeks prior to screening.
21. Poor peripheral venous access.
22. Subjects with exposure to significant diagnostic or therapeutic radiation (eg, serial X-ray, computed tomography scan, barium meal) or current employment in a job requiring radiation exposure monitoring within 12 months prior to check-in.
23. Subjects who, in the opinion of the investigator (or designee), should not participate in this study.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female subjects will be excluded to align with regulatory guidance. The 'as low as (is) reasonably achievable' (ALARA) principle prescribed by the FDA for the US recommends that radiation exposure to subjects should be kept ALARA; therefore, if no specific reason exists to include females (ie, no available data suggest metabolism of the AEF0117 is different in females versus males), then the radiation exposure to female subjects should ideally be kept at 0 by not including females in this radioactivity study and only enrolling and dosing male subjects.
Enrollment: 8 (Actual)
Dates: Start 2022-12-16 (Actual); Primary Completion 2023-02-24 (Actual); Study Completion 2023-02-24 (Actual)

PRIMARY OUTCOMES:
Urine excretion of [4-14C]AEF0117 | Up to 648 hours post dose
  Fraction excreted (Fe) based on urine collection
Feces excretion of [4-14C]AEF0117 | Up to 648 hours post dose
  Fraction excreted (Fe) based on feces collection
Area under the concentration-time curveof AEF0117 | Up to 432 hours postdose
  Area under the concentration-time curve from time 0 to the time of the last quantifiable concentration;(AUC0-t) based on serial blood sample collections and plasma AEF0117 concentration
Maximum observed concentration;of AEF0117 | Up to 432 hours postdose
  Peak Plasma Concentration (Cmax) induced by a single dose of AEF0117 will be determined based on serial blood sample collections and plasma AEF0117 concentration.
Time of the maximum observed concentration;of AEF0117 | Up to 432 hours postdose
  Time to maximum plasma concentration (tmax) of a single dose of AEF0117 will be determined based on serial blood sample collections and plasma AEF0117 concentration.
Apparent terminal elimination half-lifeof AEF0117 | Up to 432 hours postdose
  Apparent terminal elimination half-life (t1/2); based on serial blood sample collections and plasma AEF0117 concentration.
Total radioactivity | Up to 1008 hours postdose
  Measure of total radioactivity in plasma and whole blood

SECONDARY OUTCOMES:
Identification of potential metabolites | Up to 984 hours postdose
  to determine AEF0117 metabolite profiles based on plasma, urine, and feces excretion
Incidence of treatment-emergent AEs and SAEs as assessed by vital signs | 24 hours from dosing
  Evaluation by grade intensity and by evaluating changes from the baseline in vital signs
Incidence of treatment-emergent AEs and SAEs as assessed by ECGs | 24 hours from dosing
  Evaluation by grade intensity and by evaluating changes from the baseline in ECGs
Incidence of laboratory abnormalities | Up to 672 hours postdose
  Incidence of laboratory abnormalities based on hematology, clinical chemistry, and urinalysis test results

CONTACTS AND LOCATIONS:
Overall Officials: Irene Mirkin, MD, Principal Investigator — Substance Use Research Center
Locations (1):
- Labcorp Clinical Research Unit Inc., Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No